CLINICAL TRIAL: NCT01529697
Title: Prospective Study of the Feedback From an Adherence Monitor on Asthma Control
Acronym: INCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor of Medicine, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BeaumontH
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
Keywords: Asthma; Inhaler use
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Feedback (Active Comparator): In this arm patients will receive monthly review and education on inhaler technique and use based on a computer download of their last month of inhaler use
  Interventions: Behavioral: Active Feedback
- Control (Placebo Comparator): In this arm patients will be reviewed monthly, however will not have information from INCA device to tailor inhaler education.
  Interventions: Behavioral: Active Feedback

INTERVENTIONS:
Behavioral: Active Feedback — The inhaler will be fitted with a device that makes an audio recording of the inhaler use. This audio data will be downloaded to a computer program, analyzed for assessment of whether the steps involved in using the inhaler have been performed correctly. This information will be discussed with the patient.
  Other Names: Feedback from a computer log of inhaler use

SUMMARY:
Inhaled medications are the mainstay of the therapeutic management of respiratory disorders. Considered by many to be 'simple' and 'easy' to use, clinicians are aware that inhalers are often improperly used. However, there is no tool that can detect and record errors in either the timing or the method dose administration

The investigators designed a device that makes an acoustic record each time an inhaler is used. Opening the device makes an acoustic file which is recorded, this file is "time-stamped" which means that the timing of drug administration is recorded. When the device is retrieved and acoustic analysis performed, the steps involved in using the inhaler can be determined. Hence, the subjects inhaler technique is assessed and errors in the inhaler use identified. Together this means that errors in inhaler technique and timing of use can be quantified.

In this study the investigators attached the device to a discus dry powder inhaler. In order to eliminate the behavioral component of adherence and identify the mechanical issues associated with effective inhaler use the investigators studied subjects who were already in Hospital and already prescribed a discus inhaler. The investigators hypothesized that the device would identify which errors in technique were the most common and that this would provide insight into how these errors might be eliminated.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed therapy equivalent to step 3 or higher on the Asthma Management Guidelines for at least 3 months
* At least one exacerbation in the previous year with systemic glucocorticoids
* Uncontrolled/Partially Controlled Asthma by GINA guidelines

Exclusion Criteria:

* Allergy to salmeterol/fluticasone
* Patients Controlled by GINA guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adherence rate | at three months
  The rate of actual adherence at baseline and at the end of the study, which at the end of the 3 month of study will be assessed. The actual inhaler adherence, expressed as cumulative drug exposure, is calculated by combining the time of use along with the interval between doses (correct time is twice a day, in a period not less than 6 hours between the last dose and the subsequent dose or at a time greater than 18 hours apart from the previous dose.) and incorporating, by audio analysis, if the inhaler was used correctly.

SECONDARY OUTCOMES:
Asthma quality of life score | at 3 months
  The asthma quality of life score will be related to adherence, The baseline asthma quality of life score and the quality of life score at the end of three months will be subtracted and these will be correlated with the average rate of adherence over the three months.
Peak Expiratory Flow Rate | at 3 months
  The peak expiratory flow rate will be related to adherence, The baseline peak expiratory flow rate and the peak expiratory flow rate at the end of three months will be subtracted and these will be correlated with the average rate of adherence over the three months.
Asthma Control Test | at 3 months
  The asthma control test score will be related to adherence, The baseline asthma control test score and the score at the end of three months will be subtracted and these will be correlated with the average rate of adherence over the three months.
Asthma Exacerbations | over 3 months
  The frequency in exacerbations over the three months will be compared between the active and control arms.
Asthma Reliever Medication Use | over 3 months
  The change in frequency of reliever use per month from baseline to the end of the study will be compared between active and control patients.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Costello, MD, Principal Investigator — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Dublin, Ireland

REFERENCES:
- [Derived] Chan A, De Simoni A, Wileman V, Holliday L, Newby CJ, Chisari C, Ali S, Zhu N, Padakanti P, Pinprachanan V, Ting V, Griffiths CJ. Digital interventions to improve adherence to maintenance medication in asthma. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD013030. doi: 10.1002/14651858.CD013030.pub2. PMID 35691614
- [Derived] Sulaiman I, Greene G, MacHale E, Seheult J, Mokoka M, D'Arcy S, Taylor T, Murphy DM, Hunt E, Lane SJ, Diette GB, FitzGerald JM, Boland F, Sartini Bhreathnach A, Cushen B, Reilly RB, Doyle F, Costello RW. A randomised clinical trial of feedback on inhaler adherence and technique in patients with severe uncontrolled asthma. Eur Respir J. 2018 Jan 4;51(1):1701126. doi: 10.1183/13993003.01126-2017. Print 2018 Jan. PMID 29301919
- [Derived] Sulaiman I, Seheult J, MacHale E, Boland F, O'Dwyer SM, Rapcan V, D'Arcy S, Cushen B, Mokoka M, Killane I, Ryder SA, Reilly RB, Costello RW. A Method to Calculate Adherence to Inhaled Therapy that Reflects the Changes in Clinical Features of Asthma. Ann Am Thorac Soc. 2016 Nov;13(11):1894-1903. doi: 10.1513/AnnalsATS.201603-222OC. PMID 27467125
- [Derived] Sulaiman I, Mac Hale E, Holmes M, Hughes C, D'Arcy S, Taylor T, Rapcan V, Doyle F, Breathnach A, Seheult J, Murphy D, Hunt E, Lane SJ, Sahadevan A, Crispino G, Diette G, Killane I, Reilly RB, Costello RW. A protocol for a randomised clinical trial of the effect of providing feedback on inhaler technique and adherence from an electronic device in patients with poorly controlled severe asthma. BMJ Open. 2016 Jan 4;6(1):e009350. doi: 10.1136/bmjopen-2015-009350. PMID 26729384